CLINICAL TRIAL: NCT02230475
Title: Systemic Mechanisms in Allergic Rhinitis: Assessment of Metabolomic Outcomes Using the Environmental Exposure Unit (EEU). Part 2.
Brief Title: Systemic Mechanisms in Allergic Rhinitis: Assessment of Metabolomic Outcomes.
Acronym: NMR
Status: Completed | Type: Observational
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Anne Ellis, Dr. Anne K. Ellis MD MSc FRCPC, Queen's University
Other Study IDs: Kingston General Hospital
Record Dates: First submitted 2014-08-15; First posted 2014-09-03 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis; NMR
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Urine samples will be retained for analysis via nuclear magnetic resonance. Blood samples will be retained after separating the mononuclear layer. These samples will be tested for epigenetic changes. Blood samples will also be retained for IgE testing.
Oversight: Data Monitoring Committee: No

SUMMARY:
This clinical study will use the Environmental Exposure Unit (EEU) to generate allergic rhinitis symptoms in participants under controlled conditions, to collect well-characterized biological samples (urine and blood) before and after they develop these symptoms. The EEU provides the ability to control the timing, duration and levels of allergen exposure, and also other outside environmental factors, yielding ideal biologic samples for analysis with novel, cutting-edge molecular techniques. Results from the analysis of these unique allergic rhinitis samples should help determine if the technique of urine Nuclear Magnetic Resonance analysis could be a useful diagnostic tool in allergic rhinitis. IgE testing will be done on blood samples and compared to spin prick testing and symptoms of allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a healthy, ambulatory male or female volunteer 18 to 55 years of age.
* Participant has a history of Seasonal Allergic Rhinitis due to ragweed for the last two consecutive ragweed seasons.
* Participant has a positive response (wheal diameter greater than or equal to 3 mm larger than diluent control) to a skin prick test to short ragweed allergen at screening or within 12 months of screening visit.

Exclusion Criteria:

* Participant is a female that is pregnant, lactating or actively trying to become pregnant.
* smokers
* Participant is unable to comply with the washout periods for prohibited medications.
* Participant is currently receiving allergen specific immunotherapy injections.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy males and females 18-55 years old with ragweed induced allergic rhinitis.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Metabolomics | Participant visits from July 2014 - September 2014; samples and data will be analyzed and presented for up to 2 years following participant visits.
  Determine if urine NMR metabolic profiles from participants with allergic rhinitis will be significantly different from that of healthy participants (healthy controls were included in part 1 of the 2010 study) and if changes in urine NMR profile correlate with disease severity. NMR will be reported

SECONDARY OUTCOMES:
IgE testing | Participant visits from July 2014 - September 2014; samples and data will be analyzed and presented for up to 2 years following participant visits.
  Blood samples will be collected from participants to measure ragweed specific IgE levels and compare them to their individual skin testing wheal size as well as their symptoms of allergic rhinitis in the EEU before and after pollen exposure. These symptoms are reported on a questionnaire completed by the participant every 20 minutes.
Epigenetics | Participant visits from July 2014 - September 2014; samples and data will be analyzed and presented for up to 2 years following participant visits.
  Blood samples will be collected to examine epigenetic biomarkers in relation to symptoms of allergic rhinitis before and after exposure in the EEU. These symptoms are reported on a questionnaire completed by the participant every 20 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Anne K Ellis, MD MSc FRCPC, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

REFERENCES:
- See also: Related Info — http://eeu.on.ca